CLINICAL TRIAL: NCT00209274
Title: Pivotal Study: A Study of the Evalve Cardiovascular Valve Repair System - Endovascular Valve Edge-to-Edge REpair STudy (EVERESTIIRCT)
Brief Title: Pivotal Study of a Percutaneous Mitral Valve Repair System
Acronym: EVERESTIIRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #0401; Protocol #0401
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency
Keywords: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency; Mitral Valve; MR; Mitral Valve Prolapse; Edge to Edge (E2E); Alfieri Technique; MitraClip; Functional MR; Degenerative MR; Echocardiogram; CAD - Coronary Artery Disease; Heart Failure; Heart Attack; EVEREST; EVEREST I; EVEREST II; REALISM
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Coronary Artery Disease; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Percutaneous mitral valve repair using MitraClip implant. The calculated sample size was 186 patients in the device arm
  Interventions: Device: Percutaneous mitral valve repair using MitraClip implant
- 2 (Active Comparator): Mitral valve repair or replacement surgery. The calculated sample size was 93 patients in the control arm.
  Interventions: Procedure: Mitral valve repair or replacement surgery

INTERVENTIONS:
Device: Percutaneous mitral valve repair using MitraClip implant — MitraClip Implant
  Other Names: MitraClip
  Arms: 1
Procedure: Mitral valve repair or replacement surgery — Repair or replacement of mitral valve
  Arms: 2

SUMMARY:
EVEREST II Randomized Controlled Trial (RCT) is a prospective, multi-center, randomized study of the MitraClip® System in the treatment of mitral valve regurgitation, randomizing patients to MitraClip or mitral valve surgery. The EVEREST II High Risk Registry (HRR) study is a prospective multi-center study of the MitraClip System for the treatment of mitral valve regurgitation in high surgical risk patients. Enrollment in the RCT and HRR is closed. A continued access prospective, multi-center study (REALISM) of the MitraClip System in a surgical population (non-high risk arm) and a high surgical risk population (high risk arm) is ongoing. Enrollment in the non-high risk arm of REALISM is closed. Enrollment in the high risk arm of REALISM is ongoing. Patients enrolled in EVEREST II undergo 30-day, 6-month, 12-month, 18-month and 24-month clinical and echocardiographic follow-up, and then annually for 5 years.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized study of the safety and effectiveness of an endovascular approach to the treatment of mitral valve regurgitation using the Evalve Cardiovascular Valve Repair System (MitraClip® implant).

A minimum of 279 evaluable patients randomized 2:1 to MitraClip or mitral valve surgery, respectively, are required to test the primary safety and effectiveness endpoints of the RCT. Enrollment in the RCT is now complete. 60 roll-in patients were enrolled under EVEREST II RCT.

38 clinical sites throughout the US and Canada have participated in the RCT and HRR. 37 US sites are participating in REALISM.

The RCT is powered to test the hypothesis MitraClip has both superiority of safety and non-inferiority of effectiveness compared to mitral valve repair or replacement surgery. The HRR is powered to show lower mortality at 30 days with the MitraClip than predicted surgical mortality.

ELIGIBILITY:
Key Inclusion/Exclusion Criteria:

Patients with Grade 3 (moderate to severe) or Grade 4 (severe) mitral regurgitation (MR) based on American Society of Echocardiography guidelines:

* Are 18 years or older.
* Symptomatic
* If asymptomatic, must have new onset of atrial fibrillation, pulmonary hypertension, or evidence of left ventricular dysfunction
* Are candidates for mitral valve surgery
* Are candidates for transseptal catheterization
* Primary regurgitant jet must originate from malcoaptation of the A2 and P2 scallops of the mitral valve
* Appropriate valve anatomy for MitraClip
* Does not need other cardiac surgery or any emergency surgery
* Did not experience myocardial infarction in prior 12 weeks or endovascular procedure in prior 30 days
* Mitral valve orifice area ≥ 4 cm2
* Do not have renal insufficiency
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2005-08; Primary Completion 2009-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Feldman, M.D., Principal Investigator — Endeavor Health; Donald G Glower Jr., MD, Principal Investigator — Duke University Medical Center, Department of Surgery
Locations (1):
- Evanston Northwestern Healthcare, Evanston, Illinois, United States

REFERENCES:
- [Background] Fann JI, St Goar FG, Komtebedde J, Oz MC, Block PC, Foster E, Butany J, Feldman T, Burdon TA. Beating heart catheter-based edge-to-edge mitral valve procedure in a porcine model: efficacy and healing response. Circulation. 2004 Aug 24;110(8):988-93. doi: 10.1161/01.CIR.0000139855.12616.15. Epub 2004 Aug 9. PMID 15302782
- [Background] St Goar FG, Fann JI, Komtebedde J, Foster E, Oz MC, Fogarty TJ, Feldman T, Block PC. Endovascular edge-to-edge mitral valve repair: short-term results in a porcine model. Circulation. 2003 Oct 21;108(16):1990-3. doi: 10.1161/01.CIR.0000096052.78331.CA. Epub 2003 Oct 6. PMID 14530193
- [Background] Borgia F, Di Mario C, Franzen O. Adenosine-induced asystole to facilitate MitraClip placement in a patient with adverse mitral valve morphology. Heart. 2011 May;97(10):864. doi: 10.1136/hrt.2010.208132. Epub 2010 Oct 29. No abstract available. PMID 21036802
- [Background] Tamburino C, Imme S, Barbanti M, Mule M, Pistritto AM, Aruta P, Cammalleri V, Scarabelli M, Mangiafico S, Scandura S, Ussia GP. Reduction of mitral valve regurgitation with Mitraclip(R) percutaneous system. Minerva Cardioangiol. 2010 Oct;58(5):589-98. PMID 20948505
- [Background] Lim DS, Kunjummen BJ, Smalling R. Mitral valve repair with the MitraClip device after prior surgical mitral annuloplasty. Catheter Cardiovasc Interv. 2010 Sep 1;76(3):455-9. doi: 10.1002/ccd.22547. PMID 20839359
- [Background] Tamburino C, Ussia GP, Maisano F, Capodanno D, La Canna G, Scandura S, Colombo A, Giacomini A, Michev I, Mangiafico S, Cammalleri V, Barbanti M, Alfieri O. Percutaneous mitral valve repair with the MitraClip system: acute results from a real world setting. Eur Heart J. 2010 Jun;31(11):1382-9. doi: 10.1093/eurheartj/ehq051. Epub 2010 Mar 18. PMID 20299349
- [Background] Argenziano M, Skipper E, Heimansohn D, Letsou GV, Woo YJ, Kron I, Alexander J, Cleveland J, Kong B, Davidson M, Vassiliades T, Krieger K, Sako E, Tibi P, Galloway A, Foster E, Feldman T, Glower D; EVEREST Investigators. Surgical revision after percutaneous mitral repair with the MitraClip device. Ann Thorac Surg. 2010 Jan;89(1):72-80; discussion p 80. doi: 10.1016/j.athoracsur.2009.08.063. PMID 20103209
- [Background] Rogers JH, Yeo KK, Carroll JD, Cleveland J, Reece TB, Gillinov AM, Rodriguez L, Whitlow P, Woo YJ, Herrmann HC, Young JN. Late surgical mitral valve repair after percutaneous repair with the MitraClip system. J Card Surg. 2009 Nov-Dec;24(6):677-81. doi: 10.1111/j.1540-8191.2009.00901.x. Epub 2009 Jul 24. PMID 19682161
- [Background] Feldman T, Kar S, Rinaldi M, Fail P, Hermiller J, Smalling R, Whitlow PL, Gray W, Low R, Herrmann HC, Lim S, Foster E, Glower D; EVEREST Investigators. Percutaneous mitral repair with the MitraClip system: safety and midterm durability in the initial EVEREST (Endovascular Valve Edge-to-Edge REpair Study) cohort. J Am Coll Cardiol. 2009 Aug 18;54(8):686-94. doi: 10.1016/j.jacc.2009.03.077. PMID 19679246
- [Background] Herrmann HC, Kar S, Siegel R, Fail P, Loghin C, Lim S, Hahn R, Rogers JH, Bommer WJ, Wang A, Berke A, Lerakis S, Kramer P, Wong SC, Foster E, Glower D, Feldman T; EVEREST Investigators. Effect of percutaneous mitral repair with the MitraClip device on mitral valve area and gradient. EuroIntervention. 2009 Jan;4(4):437-42. doi: 10.4244/eijv4i4a76. PMID 19284064
- [Background] Luk A, Butany J, Ahn E, Fann JI, St Goar F, Thornton T, McDermott L, Madayag C, Komtebedde J. Mitral repair with the Evalve MitraClip device: histopathologic findings in the porcine model. Cardiovasc Pathol. 2009 Sep-Oct;18(5):279-85. doi: 10.1016/j.carpath.2008.07.001. Epub 2008 Aug 13. PMID 18703359
- [Background] Pope NH, Lim S, Ailawadi G. Late calcific mitral stenosis after MitraClip procedure in a dialysis-dependent patient. Ann Thorac Surg. 2013 May;95(5):e113-4. doi: 10.1016/j.athoracsur.2012.10.067. PMID 23608290
- [Background] Cikirikcioglu M, Cherian S, Schussler O, Kalangos A. Regarding "The EVEREST II Trial: design and rationale for a randomized study of the Evalve MitraClip system compared with mitral valve surgery for mitral regurgitation". Am Heart J. 2011 Jul;162(1):e11-2; author reply e13. doi: 10.1016/j.ahj.2011.04.004. Epub 2011 Jun 12. No abstract available. PMID 21742074
- [Background] Condado JA, Velez-Gimon M. Catheter-based approach to mitral regurgitation. J Interv Cardiol. 2003 Dec;16(6):523-34. doi: 10.1046/j.1540-8183.2003.01052.x. PMID 14632950
- [Background] Fann JI, St Goar FG. Percutaneous aortic valve replacement and mitral valve repair. Future Cardiol. 2005 May;1(3):393-403. doi: 10.1517/14796678.1.3.393. PMID 19804122
- [Background] Cohn LH. Percutaneous mitral valve repair with the edge-to-edge technique: a surgeon's perspective. J Am Coll Cardiol. 2005 Dec 6;46(11):2141-2. doi: 10.1016/j.jacc.2005.09.021. Epub 2005 Oct 17. No abstract available. PMID 16325054
- [Background] Condado JA, Acquatella H, Rodriguez L, Whitlow P, Velez-Gimo M, St Goar FG. Percutaneous edge-to-edge mitral valve repair: 2-year follow-up in the first human case. Catheter Cardiovasc Interv. 2006 Feb;67(2):323-5. doi: 10.1002/ccd.20603. PMID 16419054
- [Background] Feldman T, Glower D. Patient selection for percutaneous mitral valve repair: insight from early clinical trial applications. Nat Clin Pract Cardiovasc Med. 2008 Feb;5(2):84-90. doi: 10.1038/ncpcardio1068. PMID 18223540
- [Background] Biner S, Siegel RJ, Feldman T, Rafique AM, Trento A, Whitlow P, Rogers J, Moon M, Lindman B, Zajarias A, Glower D, Kar S; EVEREST investigators. Acute effect of percutaneous MitraClip therapy in patients with haemodynamic decompensation. Eur J Heart Fail. 2012 Aug;14(8):939-45. doi: 10.1093/eurjhf/hfs069. Epub 2012 May 14. PMID 22588322
- [Result] Dang NC, Aboodi MS, Sakaguchi T, Wasserman HS, Argenziano M, Cosgrove DM, Rosengart TK, Feldman T, Block PC, Oz MC. Surgical revision after percutaneous mitral valve repair with a clip: initial multicenter experience. Ann Thorac Surg. 2005 Dec;80(6):2338-42. doi: 10.1016/j.athoracsur.2005.05.030. PMID 16305903
- [Result] Feldman T, Wasserman HS, Herrmann HC, Gray W, Block PC, Whitlow P, St Goar F, Rodriguez L, Silvestry F, Schwartz A, Sanborn TA, Condado JA, Foster E. Percutaneous mitral valve repair using the edge-to-edge technique: six-month results of the EVEREST Phase I Clinical Trial. J Am Coll Cardiol. 2005 Dec 6;46(11):2134-40. doi: 10.1016/j.jacc.2005.07.065. Epub 2005 Oct 19. PMID 16325053
- [Result] Herrmann HC, Rohatgi S, Wasserman HS, Block P, Gray W, Hamilton A, Zunamon A, Homma S, Di Tullio MR, Kraybill K, Merlino J, Martin R, Rodriguez L, Stewart WJ, Whitlow P, Wiegers SE, Silvestry FE, Foster E, Feldman T. Mitral valve hemodynamic effects of percutaneous edge-to-edge repair with the MitraClip device for mitral regurgitation. Catheter Cardiovasc Interv. 2006 Dec;68(6):821-8. doi: 10.1002/ccd.20917. PMID 17080467
- [Result] Silvestry FE, Rodriguez LL, Herrmann HC, Rohatgi S, Weiss SJ, Stewart WJ, Homma S, Goyal N, Pulerwitz T, Zunamon A, Hamilton A, Merlino J, Martin R, Krabill K, Block PC, Whitlow P, Tuzcu EM, Kapadia S, Gray WA, Reisman M, Wasserman H, Schwartz A, Foster E, Feldman T, Wiegers SE. Echocardiographic guidance and assessment of percutaneous repair for mitral regurgitation with the Evalve MitraClip: lessons learned from EVEREST I. J Am Soc Echocardiogr. 2007 Oct;20(10):1131-40. doi: 10.1016/j.echo.2007.02.003. Epub 2007 Jun 13. PMID 17570634
- [Result] Mauri L, Garg P, Massaro JM, Foster E, Glower D, Mehoudar P, Powell F, Komtebedde J, McDermott E, Feldman T. The EVEREST II Trial: design and rationale for a randomized study of the evalve mitraclip system compared with mitral valve surgery for mitral regurgitation. Am Heart J. 2010 Jul;160(1):23-9. doi: 10.1016/j.ahj.2010.04.009. PMID 20598968
- [Result] Whitlow PL, Feldman T, Pedersen WR, Lim DS, Kipperman R, Smalling R, Bajwa T, Herrmann HC, Lasala J, Maddux JT, Tuzcu M, Kapadia S, Trento A, Siegel RJ, Foster E, Glower D, Mauri L, Kar S; EVEREST II Investigators. Acute and 12-month results with catheter-based mitral valve leaflet repair: the EVEREST II (Endovascular Valve Edge-to-Edge Repair) High Risk Study. J Am Coll Cardiol. 2012 Jan 10;59(2):130-9. doi: 10.1016/j.jacc.2011.08.067. PMID 22222076
- [Result] Herrmann HC, Gertz ZM, Silvestry FE, Wiegers SE, Woo YJ, Hermiller J, Segar D, Heimansohn D, Gray W, Homma S, Argenziano M, Wang A, Jollis J, Lampert MB, Alexander J, Mauri L, Foster E, Glower D, Feldman T. Effects of atrial fibrillation on treatment of mitral regurgitation in the EVEREST II (Endovascular Valve Edge-to-Edge Repair Study) randomized trial. J Am Coll Cardiol. 2012 Apr 3;59(14):1312-9. doi: 10.1016/j.jacc.2011.12.023. PMID 22464260
- [Result] Glower D, Ailawadi G, Argenziano M, Mack M, Trento A, Wang A, Lim DS, Gray W, Grayburn P, Dent J, Gillam L, Sethuraman B, Feldman T, Foster E, Mauri L, Kron I; EVEREST II Investigators. EVEREST II randomized clinical trial: predictors of mitral valve replacement in de novo surgery or after the MitraClip procedure. J Thorac Cardiovasc Surg. 2012 Apr;143(4 Suppl):S60-3. doi: 10.1016/j.jtcvs.2012.01.047. PMID 22423604
- [Result] Smith T, McGinty P, Bommer W, Low RI, Lim S, Fail P, Rogers JH. Prevalence and echocardiographic features of iatrogenic atrial septal defect after catheter-based mitral valve repair with the MitraClip system. Catheter Cardiovasc Interv. 2012 Oct 1;80(4):678-85. doi: 10.1002/ccd.23485. Epub 2012 Mar 15. PMID 22422577
- [Result] Mauri L, Foster E, Glower DD, Apruzzese P, Massaro JM, Herrmann HC, Hermiller J, Gray W, Wang A, Pedersen WR, Bajwa T, Lasala J, Low R, Grayburn P, Feldman T; EVEREST II Investigators. 4-year results of a randomized controlled trial of percutaneous repair versus surgery for mitral regurgitation. J Am Coll Cardiol. 2013 Jul 23;62(4):317-28. doi: 10.1016/j.jacc.2013.04.030. Epub 2013 May 9. PMID 23665364
- [Result] Foster E, Kwan D, Feldman T, Weissman NJ, Grayburn PA, Schwartz A, Rogers JH, Kar S, Rinaldi MJ, Fail PS, Hermiller J, Whitlow PL, Herrmann HC, Lim DS, Glower DD; EVEREST Investigators. Percutaneous mitral valve repair in the initial EVEREST cohort: evidence of reverse left ventricular remodeling. Circ Cardiovasc Imaging. 2013 Jul;6(4):522-30. doi: 10.1161/CIRCIMAGING.112.000098. Epub 2013 Apr 30. PMID 23633132
- [Derived] Ailawadi G, Lim DS, Mack MJ, Trento A, Kar S, Grayburn PA, Glower DD, Wang A, Foster E, Qasim A, Weissman NJ, Ellis J, Crosson L, Fan F, Kron IL, Pearson PJ, Feldman T; EVEREST II Investigators. One-Year Outcomes After MitraClip for Functional Mitral Regurgitation. Circulation. 2019 Jan 2;139(1):37-47. doi: 10.1161/CIRCULATIONAHA.117.031733. PMID 30586701
- [Derived] Gucuk Ipek E, Singh S, Viloria E, Feldman T, Grayburn P, Foster E, Qasim A. Impact of the MitraClip Procedure on Left Atrial Strain and Strain Rate. Circ Cardiovasc Imaging. 2018 Mar;11(3):e006553. doi: 10.1161/CIRCIMAGING.117.006553. PMID 29535132
- [Derived] Feldman T, Kar S, Elmariah S, Smart SC, Trento A, Siegel RJ, Apruzzese P, Fail P, Rinaldi MJ, Smalling RW, Hermiller JB, Heimansohn D, Gray WA, Grayburn PA, Mack MJ, Lim DS, Ailawadi G, Herrmann HC, Acker MA, Silvestry FE, Foster E, Wang A, Glower DD, Mauri L; EVEREST II Investigators. Randomized Comparison of Percutaneous Repair and Surgery for Mitral Regurgitation: 5-Year Results of EVEREST II. J Am Coll Cardiol. 2015 Dec 29;66(25):2844-2854. doi: 10.1016/j.jacc.2015.10.018. PMID 26718672
- [Derived] Wang A, Sangli C, Lim S, Ailawadi G, Kar S, Herrmann HC, Grayburn P, Foster E, Weissman NJ, Glower D, Feldman T. Evaluation of renal function before and after percutaneous mitral valve repair. Circ Cardiovasc Interv. 2015 Jan;8(1):e001349. doi: 10.1161/CIRCINTERVENTIONS.113.001349. PMID 25593120
- [Derived] Glower DD, Kar S, Trento A, Lim DS, Bajwa T, Quesada R, Whitlow PL, Rinaldi MJ, Grayburn P, Mack MJ, Mauri L, McCarthy PM, Feldman T. Percutaneous mitral valve repair for mitral regurgitation in high-risk patients: results of the EVEREST II study. J Am Coll Cardiol. 2014 Jul 15;64(2):172-81. doi: 10.1016/j.jacc.2013.12.062. PMID 25011722
- [Derived] Grayburn PA, Foster E, Sangli C, Weissman NJ, Massaro J, Glower DG, Feldman T, Mauri L. Relationship between the magnitude of reduction in mitral regurgitation severity and left ventricular and left atrial reverse remodeling after MitraClip therapy. Circulation. 2013 Oct 8;128(15):1667-74. doi: 10.1161/CIRCULATIONAHA.112.001039. Epub 2013 Sep 6. PMID 24014834
- [Derived] Siegel RJ, Biner S, Rafique AM, Rinaldi M, Lim S, Fail P, Hermiller J, Smalling R, Whitlow PL, Herrmann HC, Foster E, Feldman T, Glower D, Kar S; EVEREST Investigators. The acute hemodynamic effects of MitraClip therapy. J Am Coll Cardiol. 2011 Apr 19;57(16):1658-65. doi: 10.1016/j.jacc.2010.11.043. PMID 21492763
- [Derived] Feldman T, Foster E, Glower DD, Kar S, Rinaldi MJ, Fail PS, Smalling RW, Siegel R, Rose GA, Engeron E, Loghin C, Trento A, Skipper ER, Fudge T, Letsou GV, Massaro JM, Mauri L; EVEREST II Investigators. Percutaneous repair or surgery for mitral regurgitation. N Engl J Med. 2011 Apr 14;364(15):1395-406. doi: 10.1056/NEJMoa1009355. Epub 2011 Apr 4. PMID 21463154
- [Derived] Ladich E, Michaels MB, Jones RM, McDermott E, Coleman L, Komtebedde J, Glower D, Argenziano M, Feldman T, Nakano M, Virmani R; Endovascular Valve Edge-to-Edge Repair Study (EVEREST) Investigators. Pathological healing response of explanted MitraClip devices. Circulation. 2011 Apr 5;123(13):1418-27. doi: 10.1161/CIRCULATIONAHA.110.978130. Epub 2011 Mar 21. PMID 21422390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The EVEREST II RCT was conducted in patients who were indicated for and could undergo mitral valve surgery. A total of 279 patients were enrolled at United States & Canada investigational sites between Aug 5,2005 to Sep 17,2008 time period. The subjects were randomized to Device group (n=184; MitraClip) &Control group (n=95;Mitral Valve Surgery).
Pre-assignment Details: The EVEREST II RCT enrolled 279 patients (184 Device and 95 Control), of whom 21 patients (6 Device and 15 Control) did not undergo treatment per their randomized assignment, and are reported as "randomized not treated" (RNT). All RNT patients except one withdrew from the trial.
Groups:
- Device Group (MitraClip Device): Percutaneous mitral valve repair using MitraClip implant.
- Control Group (Mitral Valve Surgery): Mitral valve repair or replacement surgery.
Period: Overall Study
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Started | 184 | 95
Completed | 113 | 48
Not Completed | 71 | 47
Not completed — Missed visit | 3 | 2
Not completed — Death | 32 | 15
Not completed — Withdrawal by Subject | 30 | 15
Not completed — Randomized not treated (RNT) | 6 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery) | Total
Number analyzed (Participants) | 184 | 95 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (12.8) | 65.7 (12.9) | 66.7 (12.8)
Age, Customized [Count of Participants; unit: Participants]
  18-75 years | 129 | 69 | 198
  >75 years | 55 | 26 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 32 | 101
  Male | 115 | 63 | 178
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 177 | 93 | 270
  Canada | 7 | 2 | 9
NYHA Functional Class [Count of Participants; unit: Participants] — Class I: Patients with cardiac disease but without resulting limitations of physical activity. Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or anginal syndrome may be present even at rest & discomfort is increased with physical activity.
  Participants
    NYHA Functional Class I | 17 | 19 | 36
    NYHA Functional Class II | 73 | 31 | 104
    NYHA Functional Class III | 82 | 41 | 123
    NYHA Functional Class IV | 12 | 4 | 16
Mitral regurgitation (MR) [Count of Participants; unit: Participants]
  0: None | 0 | 0 | 0
  1+: Mild | 0 | 0 | 0
  2+: Moderate | 8 | 7 | 15
  3+: Moderate-to-Severe | 130 | 67 | 197
  4+: Severe | 46 | 21 | 67
Left Ventricular (LV) Measurement [Mean (Standard Deviation); unit: mL]
  LV End Diastolic Volume (LVEDV) | 156.5 (39.0) | 159.6 (46.3) | 158.05 (42.65)
  LV End Systolic Volume (LVESV) | 63.5 (25.5) | 63.8 (28.9) | 63.65 (27.20)
Left Ventricular (LV) Measurement [Mean (Standard Deviation); unit: cm]
  LV internal dimension diastole (LVIDd) | 5.5 (0.7) | 5.5 (0.7) | 5.5 (0.7)
  LV internal dimension systole (LVIDs) | 3.7 (0.9) | 3.5 (0.8) | 3.6 (0.85)
36-Item Short Form Health Survey (SF-36) Quality of Life (QOL) [Mean (Standard Deviation); unit: scores on a scale] — The SF-36 is a multidimensional, patient-reported survey containing 36 questions on a 0-100 scale measuring physical (Physical Component Score PCS) & mental health status (Mental Component Score MCS) in relation to 8 health concepts: physical functioning, role limitations due to physical or emotional health, bodily pain, general health perceptions, vitality, social functioning, & general mental health. Higher scores represent better self-perceived health. The PCS & MCS norms for 65-75 year olds are 44 and 52, while the norms for CHF population are 31 and 46, respectively.
  scores on a scale
    Physical Component Score | 41.1 (10.0) | 41.9 (11.1) | 41.4 (10.3)
    Mental Component Score | 47.1 (11.9) | 46.6 (12.5) | 46.9 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: Defined as a combined clinical endpoint of death, myocardial infarction, reoperation for failed surgical repair or replacement, nonelective cardiovascular surgery for adverse events, stroke, renal failure, deep wound infection, ventilation for greater than 48 hours, gastrointestinal (GI) complication requiring surgery, new onset of permanent atrial fibrillation, septicemia, and transfusion of 2 or more units of blood.
Time Frame: 30 days
Population: Per-protocol cohort. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 136 | 79
Participants | 13 | 45

2. Primary Outcome: Number of Participants With Freedom From Surgery for Valve Dysfunction, Death, and Moderate to Severe (3+) or Severe (4+) Mitral Regurgitation (MR).
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 134 | 74
Participants | 97 | 65

3. Secondary Outcome: Freedom From All-Cause Mortality
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 70
Percentage of participants | 93.7 | 92.3

4. Secondary Outcome: Freedom From All-Cause Mortality
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 143 | 65
Percentage of participants | 90.0 | 89.6

5. Secondary Outcome: Freedom From All-Cause Mortality
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 133 | 57
Percentage of participants | 87.5 | 85.3

6. Secondary Outcome: Freedom From All-Cause Mortality
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 119 | 52
Percentage of participants | 83.4 | 82.3

7. Secondary Outcome: Freedom From All-Cause Mortality
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 58 | 24
Percentage of participants | 81.2 | 79

8. Secondary Outcome: Number of Participants With Freedom From Surgery for Valve Dysfunction, Death, and Moderate to Severe (3+) or Severe (4+) Mitral Regurgitation.
Time Frame: 12 months
Population: Intent-to-treat (ITT) population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 175 | 89
Participants | 118 | 65

9. Secondary Outcome: Number of Participants With Freedom From Surgery for Valve Dysfunction, Death, and Moderate to Severe (3+) or Severe (4+) Mitral Regurgitation (MR).
Time Frame: 24 months
Population: Per-protocol population.The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 126 | 68
Participants | 87 | 55

10. Secondary Outcome: Number of Participants With Freedom From Surgery for Valve Dysfunction, Death, and Moderate to Severe (3+) or Severe (4+) Mitral Regurgitation (MR) in Intention to Treat Strategy Cohort
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 161 | 83
participants | 100 | 56

11. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as determined by the core echo laboratory at 30 days or hospital discharge, whichever is longer.
Time Frame: At discharge (≤ 14 days following index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of volume ejected
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 170 | 77
Percentage of volume ejected | 56.9 (10.0) | 53.9 (10.9)

12. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as determined by the core echo laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of volume ejected
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 144 | 65
Percentage of volume ejected | 58.0 (8.7) | 55.3 (10.2)

13. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as determined by the core echo laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of volume ejected
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 125 | 56
Percentage of volume ejected | 56.9 (8.3) | 55.8 (8.1)

14. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as determined by the core echo laboratory.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of volume ejected
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 119 | 47
Percentage of volume ejected | 57.0 (9.1) | 58.4 (9.2)

15. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as determined by the core echo laboratory.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of volume ejected
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 102 | 45
Percentage of volume ejected | 57.6 (9.9) | 58.9 (10.2)

16. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF as determined by the core echo laboratory.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of volume ejected
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 105 | 40
Percentage of volume ejected | 56.5 (10.1) | 57 (9.3)

17. Secondary Outcome: Left Ventricular Status- Left Ventricular End-diastolic Volume (LVEDV), Left Ventricular End-systolic Volume (LVESV)
Description: Left Ventricular Status includes Left ventricular (LV) end-diastolic volume (LVEDV), LV end-systolic volume (LVESV), as determined by the core echo laboratory at 30 days or hospital discharge, whichever is longer.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 170 | 77
ml
  LVEDV | 144.7 (40.0) | 130.8 (40.5)
  LVESV | 63.7 (27.2) | 62.0 (29.2)

18. Secondary Outcome: Left Ventricular Status- LVEDV, LVESV
Description: Left Ventricular Status includes LV end-diastolic volume (LVEDV), LV end-systolic volume (LVESV),as determined by the core echo laboratory at 12 months.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 144 | 65
ml
  LVEDV | 133.7 (35.5) | 120.9 (44.3)
  LVESV | 57.5 (24.0) | 56.2 (31.4)

19. Secondary Outcome: Left Ventricular Status- LVEDV, LVESV
Description: Left Ventricular Status includes LV end-diastolic volume (LVEDV), LV end-systolic volume (LVESV), as determined by the core echo laboratory at 24 months.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 125 | 56
mL
  LVEDV | 123.4 (35.0) | 110.5 (40.9)
  LVESV | 54.7 (24.7) | 50.4 (26.3)

20. Secondary Outcome: Left Ventricular Status- LVEDV, LVESV
Description: Left Ventricular Status includes LV end-diastolic volume (LVEDV), LV end-systolic volume (LVESV), as determined by the core echo laboratory at 3 years.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 119 | 47
ml
  LVEDV | 130.6 (32.6) | 112.7 (40.2)
  LVESV | 57.7 (24.7) | 48.0 (24.7)

21. Secondary Outcome: Left Ventricular Status- LVEDV, LVESV
Description: Left Ventricular Status includes LV end-diastolic volume (LVEDV), LV end-systolic volume (LVESV), as determined by the core echo laboratory at 4 years
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 102 | 45
ml
  LVEDV | 126.6 (33.1) | 112.7 (40.4)
  LVESV | 55.0 (24.4) | 48.1 (26.9)

22. Secondary Outcome: Left Ventricular Status- LVEDV, LVESV
Description: Left Ventricular Status includes LV end-diastolic volume (LVEDV), LV end-systolic volume (LVESV), as determined by the core echo laboratory at 5 years.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 105 | 40
ml
  LVEDV | 126.3 (32.5) | 112.9 (37.8)
  LVESV | 56.1 (23) | 50.1 (26.3)

23. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Left Ventricular internal dimension systole (LVIDs) as determined by the core echo laboratory.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 169 | 77
cm | 3.6 (0.9) | 3.5 (0.8)

24. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Left Ventricular internal dimension systole (LVIDs) as determined by the core echo laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 146 | 66
cm | 3.5 (0.8) | 3.3 (0.8)

25. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Left Ventricular internal dimension systole (LVIDs) as determined by the core echo laboratory.
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 125 | 58
cm | 3.4 (0.8) | 3.2 (0.9)

26. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Left Ventricular internal dimension systole (LVIDs) as determined by the core echo laboratory.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 120 | 50
cm | 3.6 (0.9) | 3.2 (0.8)

27. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Left Ventricular internal dimension systole (LVIDs) as determined by the core echo laboratory.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 102 | 46
cm | 3.6 (0.9) | 3.3 (0.8)

28. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Left Ventricular internal dimension systole (LVIDs) as determined by the core echo laboratory.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 104 | 42
cm | 3.6 (0.9) | 3.3 (0.9)

29. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Left Ventricular internal dimension diastole (LVIDd) as determined by the core echo laboratory.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 171 | 77
cm | 5.3 (0.7) | 5.0 (0.7)

30. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Left Ventricular internal dimension diastole (LVIDd) as determined by the core echo laboratory at 12 months.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 148 | 66
cm | 5.1 (0.7) | 4.8 (0.7)

31. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Left Ventricular internal dimension diastole (LVIDd) as determined by the core echo laboratory at 24 months.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 127 | 58
cm | 5.0 (0.7) | 4.7 (0.8)

32. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Left Ventricular internal dimension diastole (LVIDd) as determined by the core echo laboratory at 3 years.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 122 | 50
cm | 5.2 (0.7) | 4.8 (0.7)

33. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Left Ventricular internal dimension diastole (LVIDd) as determined by the core echo laboratory at 4 years.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 102 | 46
cm | 5.3 (0.6) | 4.8 (0.7)

34. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Left Ventricular internal dimension diastole (LVIDd) as determined by the core echo laboratory at 5 years.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 106 | 42
cm | 5.2 (0.6) | 4.9 (0.7)

35. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: Baseline
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants
  NYHA Functional Class I | 17 | 19
  NYHA Functional Class II | 73 | 31
  NYHA Functional Class III | 82 | 41
  NYHA Functional Class IV | 12 | 4

36. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: as for outcome 35
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 168 | 75
Participants
  NYHA Functional Class I | 84 | 40
  NYHA Functional Class II | 67 | 28
  NYHA Functional Class III | 17 | 7
  NYHA Functional Class IV | 0 | 0

37. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: as for outcome 35
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 151 | 66
Participants
  NYHA Functional Class I | 104 | 46
  NYHA Functional Class II | 44 | 12
  NYHA Functional Class III | 3 | 7
  NYHA Functional Class IV | 0 | 1

38. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: as for outcome 35
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 132 | 60
Participants
  NYHA Functional Class I | 89 | 43
  NYHA Functional Class II | 42 | 11
  NYHA Functional Class III | 1 | 4
  NYHA Functional Class IV | 0 | 2

39. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: as for outcome 35
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 120 | 50
Participants
  NYHA Functional Class I | 84 | 41
  NYHA Functional Class II | 32 | 8
  NYHA Functional Class III | 4 | 1
  NYHA Functional Class IV | 0 | 0

40. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: as for outcome 35
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 105 | 48
Participants
  NYHA Functional Class I | 70 | 35
  NYHA Functional Class II | 29 | 10
  NYHA Functional Class III | 6 | 3
  NYHA Functional Class IV | 0 | 0

41. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease.
Description: as for outcome 35
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 106 | 42
Participants
  NYHA Functional Class I | 70 | 33
  NYHA Functional Class II | 27 | 8
  NYHA Functional Class III | 9 | 1
  NYHA Functional Class IV | 0 | 0

42. Secondary Outcome: New York Heart Association (NYHA) Functional Class Cardiac Disease: NYHA Functional Class III or IV
Description: as for outcome 35
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 168 | 75
Percentage of participants | 10.1 | 9.3

43. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease: NYHA Functional Class III or IV
Description: as for outcome 35
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 151 | 66
Percentage of participants | 2.0 | 12.1

44. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease: NYHA Functional Class III or IV
Description: as for outcome 35
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 132 | 60
Percentage of participants | 0.8 | 10.0

45. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease: NYHA Functional Class III or IV
Description: as for outcome 35
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 120 | 50
Percentage of participants | 3.3 | 2.0

46. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease: NYHA Functional Class III or IV
Description: as for outcome 35
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 105 | 48
Percentage of participants | 5.7 | 6.3

47. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Functional Class Cardiac Disease: NYHA Functional Class III or IV
Description: as for outcome 35
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 106 | 42
Percentage of participants | 8.5 | 2.4

48. Secondary Outcome: Short Form (SF)-36 Quality of Life Questionnaire.
Description: The SF-36 is a multidimensional, patient-reported survey containing 36 questions on a 0-100 scale measuring physical (Physical Component Score) & mental health status (Mental Component Score) in relation to 8 health concepts: physical functioning, role limitations due to physical or emotional health, bodily pain, general health perceptions, vitality, social functioning, & general mental health. Responses to each of the SF-36 items are scored and expressed as a score on a 0-100 scale (0% in a domain represents the poorest possible QOL&100% indicates full QOL).Higher scores represent better self-perceived health.
  The physical & mental functions were assessed by the Physical Component Summary (PCS) score & Mental Component Summary (MCS) score. Normal PCS and MCS scores vary depending on the demographics of the population studied. The PCS&MCS norms for 65-75 year old are 44 & 52, respectively while the norms for CHF population are 31 & 46, respectively.
Time Frame: 30 days
Population: The SF-36 questionnaire consists of 36 questions in relation to eight health concepts:
  Physical functioning, role limitations due to physical health, bodily pain,general health perceptions,vitality (energy/fatigue),social functioning,role limitations due to emotional health and general mental health (psychological distress/wellbeing).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 159 | 68
scores on a scale
  Physical Component Summary | 43.8 (9.8) | 36.9 (9.9)
  Mental Component Summary | 50.8 (10.8) | 46.7 (12.4)

49. Secondary Outcome: Short Form (SF)-36 Quality of Life Questionnaire.
Description: as for outcome 48
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 139 | 64
scores on a scale
  Physical Component Summary | 46.8 (9.5) | 46.5 (10.6)
  Mental Component Summary | 52.9 (8.0) | 50.4 (10.9)

50. Secondary Outcome: Cardiac Output
Description: Cardiac output as measured by core lab echocardiography.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 162 | 71
L/min | 4.2 (1.2) | 4.8 (1.3)

51. Secondary Outcome: Cardiac Output
Description: Cardiac output as measured by core lab echocardiography.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 147 | 67
L/min | 4.4 (1.3) | 4.6 (1.4)

52. Secondary Outcome: Cardiac Output
Description: Cardiac output as measured by core lab echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 121 | 57
L/min | 4.0 (1.1) | 4.1 (1.1)

53. Secondary Outcome: Cardiac Index
Description: Defined as cardiac output divided by body surface area, as measured by core lab echocardiography.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 71
L/min/m^2 | 2.2 (0.6) | 2.5 (0.6)

54. Secondary Outcome: Cardiac Index (CI)
Description: Defined as cardiac output divided by body surface area as measured by core lab echocardiography. CI is a normalization of cardiac output to take into account the effect of body size on cardiac output requirements.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 145 | 65
L/min/m^2 | 2.3 (0.6) | 2.4 (0.6)

55. Secondary Outcome: Cardiac Index
Description: Defined as cardiac output divided by body surface area, as measured by core lab echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 121 | 56
L/min/m^2 | 2.1 (0.5) | 2.1 (0.5)

56. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as determined by the core echo laboratory. In the presence of regurgitation of one valve, without any intracardiac shunt, the flow through the affected valve is larger than through other competent valves. The difference between the two represents the regurgitant volume.
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 131 | 45
mL | 22.7 (17.6) | 13.1 (10.7)

57. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as determined by the core echo laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 115 | 34
mL | 19.9 (14.4) | 14.6 (10.5)

58. Secondary Outcome: Regurgitant Volume
Description: Regurgitant volume as determined by the core echo laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 85 | 25
mL | 19.4 (13.2) | 15.7 (10.5)

59. Secondary Outcome: Regurgitant Fraction (RF)
Description: RF is defined as the percentage of the left ventricular (LV) stroke volume that regurgitates into the left atrium.
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of LV stroke volume
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 131 | 45
percentage of LV stroke volume | 25.4 (15.3) | 17.3 (13.1)

60. Secondary Outcome: Regurgitant Fraction
Description: Regurgitant fraction is defined as the percentage of the left ventricular (LV) stroke volume that regurgitates into the left atrium.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of LV stroke volume
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 115 | 34
Percentage of LV stroke volume | 22.8 (13.8) | 19.2 (12.1)

61. Secondary Outcome: Regurgitant Fraction
Description: as for outcome 60
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percentage of LV stroke volume
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 85 | 25
Percentage of LV stroke volume | 24.5 (13.3) | 20.4 (10.9)

62. Secondary Outcome: Number of Participants With Clip Implant Rate
Description: Defined as the rate of successful implantation of MitraClip(s).
Time Frame: Day 0
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame. MitraClip was not implanted in control group, hence overall number of patients analyzed will remain 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 0
Participants | 158 |

63. Secondary Outcome: Number of Participants With Acute Procedural Success
Description: Defined as successful MitraClip implantation with resulting MR of 2+ or less.
Time Frame: 30 Days
Population: ITT population. The number of participants analyzed in Device group includes subjects who had available follow up data at that time frame. Not applicable for Mitral valve surgery patients as device was not implanted.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 0
Participants | 137 |

64. Secondary Outcome: Number of Participants With Acute Surgical Success
Description: Defined as successful mitral valve repair or replacement surgery.
Time Frame: 30 Days
Population: The number of participants analyzed in control group includes subjects who had available follow up data at that time frame. Not applicable for Device group patients as device was not implanted. The population includes all patients who underwent the index surgical procedure and excludes 15 patients who were randomized, but not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 0 | 80
Participants |  | 80

65. Secondary Outcome: Number of Participants With Successful Clip Implant and Acute Procedural Success
Description: Acute procedural success is defined as MR severity ≤ 2 at discharge or 1 grade MR reduction at discharge accompanied by 1 level NYHA reduction.
Time Frame: 30 days
Population: The number of participants analyzed in Device group includes subjects who had available follow up data at that time frame. Not applicable for Mitral valve surgery patients as device was not implanted.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 0
Participants
  Device Implant Rate | 158 |
  Acute Procedural Success | 137 |

66. Secondary Outcome: Number of Participants With Mitral Valve Repair Success.
Description: Defined as freedom from mitral valve replacement surgery for Valve Dysfunction, death, re-operation, and MR > 2+ at 12 months.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 177 | 91
Participants | 114 | 57

67. Secondary Outcome: Number of Participants With Mitral Valve Repair Success.
Description: as for outcome 66
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 167 | 84
Participants | 103 | 46

68. Secondary Outcome: Number of Participants With Procedural Freedom From In-hospital MAE.
Time Frame: Day 0
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 168 | 41

69. Secondary Outcome: Number of Participants With Procedural Freedom From In-hospital MAE
Time Frame: Day 30
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 10 | 39

70. Secondary Outcome: Number of Participants With MAE: Surgery After Device and First Time Surgery Control
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 37 | 80
Participants | 14 | 40

71. Secondary Outcome: Number of Participants With Major Vascular Complications
Description: Vascular Complications defined as the occurrence of any of the following resulting through 30 days or hospital discharge, whichever is longer:
  * Hematoma at access site >6 cm;
  * Retroperitoneal hematoma;
  * Arteriovenous (AV) fistula;
  * Symptomatic peripheral ischemia / nerve injury or the clinical signs or symptoms lasting >48 hours;
  * Vascular Surgical Repair at catheter access sites;
  * Pulmonary embolism;
  * Ipsilateral deep vein thrombus; or
  * Access site-related infection requiring intravenous antibiotics and/or extended hospitalization.
Time Frame: 30 days
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 9 | 0

72. Secondary Outcome: Number of Participants With Major Vascular Complications
Description: as for outcome 71
Time Frame: 12 months
Population: as for outcome 71
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 11 | 0

73. Secondary Outcome: Number of Participants With Major Bleeding Complications.
Description: Major Bleeding Complications defined as procedure related bleeding that requires a transfusion of ≥2 units of blood products and/or surgical intervention at 30 days or hospital discharge, whichever is longer.
Time Frame: 30 days
Population: as for outcome 71
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 9 | 38

74. Secondary Outcome: Number of Participants With Major Bleeding Complications.
Description: Major Bleeding Complications defined as procedure related bleeding that requires a transfusion of ≥2 units of blood products and/or surgical intervention at 12 months.
Time Frame: 12 months
Population: as for outcome 71
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 17 | 39

75. Secondary Outcome: Number of Participants With Major Adverse Events (MAE)
Time Frame: 12 months.
Population: Intent to treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 39 | 44

76. Secondary Outcome: Number of Participants With MAE in Patients Over 75 Years of Age.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 55 | 26
Participants | 9 | 12

77. Secondary Outcome: Number of Participants With MAE in Patients Over 75 Years of Age.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 55 | 26
Participants | 14 | 14

78. Secondary Outcome: Number of Participants With Dysrhythmia
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 9 | 22

79. Secondary Outcome: Number of Participants With Dysrhythmia
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 22 | 22

80. Secondary Outcome: Number of Participants With Endocarditis.
Description: Defined as a diagnosis of endocarditis based on the Duke criteria. Infection in the lining of the heart, of the valves, or of the muscles of the heart. Signs of endocarditis may include persistent positive blood cultures and/or valvular structural abnormality and vegetations as seen using echocardiography.
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 1 | 1

81. Secondary Outcome: Number of Participants With Endocarditis.
Description: as for outcome 80
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 2 | 1

82. Secondary Outcome: Number of Participants With Thrombosis.
Description: Defined as evidence of the formation of an independently moving thrombus on any part of the MitraClip or any commercially available implant used during surgery by echocardiography or fluoroscopy.
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 0 | 0

83. Secondary Outcome: Number of Participants With Thrombosis.
Description: as for outcome 82
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 0 | 0

84. Secondary Outcome: Number of Participants With Hemolysis
Description: Defined as new onset of anemia associated with laboratory evidence of red cell destruction. Diagnosed when plasma free hemoglobin is greater than 40 mg/dL on repeat measures within 24 hours or on one measure if intervention is initiated based on other clinical symptoms. Reported as major or minor as defined below:
  Major: Requires intervention with red blood cell transfusion or other hematocrit increasing measures in the absence of other obvious bleeding.
  Minor: Does not require intervention.
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 0 | 0

85. Secondary Outcome: Number of Participants With Hemolysis
Description: as for outcome 84
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 0 | 0

86. Secondary Outcome: Number of Participants With Clinically Significant Atrial Septal Defect (ASD).
Description: Defined as a significant residual atrial septal opening. Reported as clinically significant if intervention is performed for the primary purpose of repairing the ASD. If cardiac surgery is indicated for reasons other than residual ASD (e.g., residual MR) and the ASD is repaired at the same time, this does not meet the definition of clinically significant ASD.
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 2 | 0

87. Secondary Outcome: Number of Participants With Clinically Significant Atrial Septal Defect (ASD)
Description: as for outcome 86
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 4 | 0

88. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Defined as a mitral valve planimetered orifice area of less than 1.5 cm^2 as measured by echocardiography.
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 0 | 0

89. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Defined as a mitral valve planimetered orifice area of less than 1.5 cm^2 as measured by echocardiography.
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 0 | 0

90. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Defined as a mitral valve planimetered orifice area of less than 1.5 cm^2 as measured by echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 0 | 1

91. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: Defined as a mitral valve (MV) planimetered orifice area of less than 1.5 cm^2 as measured by echocardiography. A "confirmed" case of MV stenosis is defined as Echocardiography Core Lab (ECL) measured mitral valve orifice area < 1.5 cm^2. A "conservative" case of MV stenosis is defined as stenosis suspected by the site, based on hemodynamic measurements or clinical symptoms.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants
  Conservative cases | 3 | 0
  Confirmed cases | 0 | 0

92. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: as for outcome 91
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants
  Conservative cases | 3 | 0
  Confirmed cases | 0 | 0

93. Secondary Outcome: Number of Participants With Mitral Valve Stenosis
Description: as for outcome 91
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants
  Conservative cases | 4 | 2
  Confirmed cases | 1 | 0

94. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: At Discharge (≤14 days of index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 140 | 59
cm^2 | 3.7 (1.4) | 3.6 (0.9)

95. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 121 | 53
cm^2 | 3.6 (1.1) | 3.9 (1.2)

96. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 100 | 47
cm^2 | 3.2 (1.0) | 3.7 (1.1)

97. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 90 | 35
cm^2 | 3.3 (0.9) | 3.3 (0.8)

98. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 81 | 34
cm^2 | 3.3 (0.9) | 3.6 (0.9)

99. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 82 | 31
cm^2 | 3.2 (0.9) | 3.8 (0.8)

100. Secondary Outcome: Mitral Valve Area by Planimetry
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 75 | 30
cm^2 | 3.2 (1.0) | 3.7 (1.0)

101. Secondary Outcome: Mitral Valve Area by Planimetry Index
Description: Defined as mitral valve area divided by body surface area as measured by core lab echocardiography.
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 118 | 53
cm^2/m^2 | 1.9 (0.6) | 2.0 (0.5)

102. Secondary Outcome: Mitral Valve Area by Planimetry Index
Description: Defined as mitral valve area divided by body surface area as measured by core lab echocardiography.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 105 | 48
cm^2/m^2 | 1.7 (0.5) | 1.9 (0.6)

103. Secondary Outcome: Mitral Valve Area by Planimetry Index
Description: Defined as mitral valve area divided by body surface area as measured by core lab echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 92 | 36
cm^2/m^2 | 1.7 (0.4) | 1.8 (0.6)

104. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: At Discharge (≤14 days of index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 166 | 71
cm^2 | 3.0 (1.1) | 3.3 (1.1)

105. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 156 | 66
cm^2 | 2.8 (1.0) | 3.5 (1.2)

106. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 140 | 63
cm^2 | 2.9 (1.0) | 3.1 (1.1)

107. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 121 | 52
cm^2 | 2.7 (0.7) | 2.8 (0.7)

108. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 120 | 48
cm^2 | 2.7 (0.7) | 2.8 (0.6)

109. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 102 | 48
cm^2 | 2.9 (0.8) | 3.0 (1.0)

110. Secondary Outcome: Mitral Valve Area by Pressure Half-time
Description: Mitral valve area as measured by core lab echocardiography.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 101 | 41
cm^2 | 2.7 (0.7) | 2.8 (0.7)

111. Secondary Outcome: Mitral Valve Area by Pressure Half-time Index
Description: Defined as mitral valve area divided by body surface area as measured by core lab echocardiography.
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 153 | 66
cm^2/m^2 | 1.5 (0.6) | 1.9 (0.7)

112. Secondary Outcome: Mitral Valve Area by Pressure Half-time Index
Description: Defined as mitral valve area divided by body surface area as measured by core lab echocardiography.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 142 | 65
cm^2/m^2 | 1.5 (0.6) | 1.7 (0.7)

113. Secondary Outcome: Mitral Valve Area by Pressure Half-time Index
Description: Defined as mitral valve area divided by body surface area as measured by core lab echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 123 | 54
cm^2/m^2 | 1.4 (0.4) | 1.5 (0.5)

114. Secondary Outcome: Transvalvular Mitral Valve Gradient
Description: Defined as the mean pressure gradient across the mitral valve as measured by echocardiography.
Time Frame: At Discharge (≤ 14 days following index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 168 | 73
mmHg | 3.3 (1.9) | 3.1 (1.6)

115. Secondary Outcome: Transvalvular Mitral Mean Pressure Gradient (Mean MVG)
Description: Defined as the mean pressure gradient across the mitral valve as measured by Echocardiography Core Laboratory (ECL).
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 140 | 64
mmHg | 3.2 (1.7) | 3.1 (1.2)

116. Secondary Outcome: Transvalvular Mitral Mean Pressure Gradient (Mean MVG)
Description: Defined as the mean pressure gradient across the mitral valve as measured by echocardiography.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 121 | 53
mmHg | 2.8 (1.4) | 2.9 (1.8)

117. Secondary Outcome: Transvalvular Mitral Mean Pressure Gradient (Mean MVG)
Description: Defined as the mean pressure gradient across the mitral valve as measured by echocardiography.
Time Frame: 3 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 120 | 48
mmHg | 3.0 (1.5) | 2.8 (1.4)

118. Secondary Outcome: Transvalvular Mitral Mean Pressure Gradient (Mean MVG)
Description: Defined as the mean pressure gradient across the mitral valve as measured by echocardiography.
Time Frame: 4 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 102 | 48
mmHg | 3.0 (1.4) | 3.1 (1.5)

119. Secondary Outcome: Transvalvular Mitral Mean Pressure Gradient (Mean MVG)
Description: Defined as the mean pressure gradient across the mitral valve as measured by echocardiography.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 104 | 41
mmHg | 3.0 (1.4) | 3.0 (1.4)

120. Secondary Outcome: Post-procedure Length of Hospital Stay
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
days | 2.6 (6.3) | 7.5 (4)

121. Secondary Outcome: Post-procedure Intensive Care Unit (ICU) / Critical Care Unit (CCU) Duration
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 176 | 77
hours | 38.6 (135.9) | 82.3 (84.9)

122. Secondary Outcome: Number of Participants With Hospital Re-admissions
Description: Defined as re-admission to the hospital for any reason. The endpoint was intended to capture each time a patient was re-admitted to the hospital for any reason and was to be reported as a rate through 30 days for both the Device and Control groups.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 171 | 76
Participants | 24 | 14

123. Secondary Outcome: Number of Participants With Incidence of Discharge to a Nursing Home or Skilled Nursing Facility/Hospital
Time Frame: 30 Days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 6 | 12

124. Secondary Outcome: Number of Participants With Incidence of Hospital Readmissions for Congestive Heart Failure (CHF).
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 171 | 76
Participants | 2 | 2

125. Secondary Outcome: Number of Participants With New Coumadin (Warfarin) Usage
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 143 | 65
Participants | 13 | 29

126. Secondary Outcome: Number of Participants With New Coumadin (Warfarin) Usage
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 143 | 65
Participants | 36 | 33

127. Secondary Outcome: Number of Participants With Durability of the MitraClip Device and Surgery.
Description: Device group: Freedom from death, surgery for mitral valve dysfunction and MR > 2+ at the end of each follow-up interval.
  Control group: Freedom from death, re-operation for mitral valve dysfunction and MR > 2+ at the end of each follow-up interval.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 137 | 80
Participants
  Deaths | 6 | 5
  Surgeries | 9 | 2
  Patients with MR > 2+ | 22 | 2
  Withdrawn/ Censored | 3 | 6

128. Secondary Outcome: Number of Participants With Durability of the MitraClip Device and Surgery.
Description: as for outcome 127
Time Frame: 12-18 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 97 | 65
Participants
  Deaths | 0 | 0
  Surgeries | 0 | 1
  Patients with MR > 2+ | 4 | 2
  Withdrawn/ Censored | 29 | 25

129. Secondary Outcome: Number of Participants With Durability of the MitraClip Device and Surgery.
Description: as for outcome 127
Time Frame: 18-24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 64 | 37
Participants
  Deaths | 0 | 0
  Surgeries | 0 | 0
  Patients with MR > 2+ | 3 | 0
  Withdrawn/ Censored | 19 | 12

130. Secondary Outcome: Number of Participants With Durability of the MitraClip Device and Surgery.
Description: as for outcome 127
Time Frame: 24 months-3 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 87 | 55
Participants
  Deaths | 0 | 2
  Surgeries | 0 | 1
  Patients with MR > 2+ | 4 | 0
  Withdrawn/ Censored | 52 | 32

131. Secondary Outcome: Number of Participants With Freedom From Death, Mitral Valve Surgery/Re-operation and MR > 2+
Description: Durability estimates: Freedom from Death, Mitral Valve Surgery/Re-operation and MR > 2+
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 110 | 71

132. Secondary Outcome: Number of Participants With Freedom From Death, Mitral Valve Surgery/Re-operation and MR > 2+
Description: Durability estimates: Freedom from Death, Mitral Valve Surgery/Re-operation and MR > 2+
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 101 | 66

133. Secondary Outcome: Number of Participants With Freedom From Death, Mitral Valve Surgery/Re-operation and MR > 2+
Description: Durability estimates: Freedom from Death, Mitral Valve Surgery/Re-operation and MR > 2+
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 96 | 62

134. Secondary Outcome: Number of Participants With Freedom From Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Mitral Valve Surgery/Re-operation
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 141 | 78

135. Secondary Outcome: Number of Participants With Freedom From Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Mitral Valve Surgery/Re-operation
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 140 | 77

136. Secondary Outcome: Number of Participants With Freedom From Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Mitral Valve Surgery/Re-operation
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 139 | 76

137. Secondary Outcome: Number of Participants With Freedom From Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Mitral Valve Surgery/Re-operation
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 137 | 76

138. Secondary Outcome: Number of Participants With Freedom From Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Mitral Valve Surgery/Re-operation
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 135 | 75

139. Secondary Outcome: Number of Participants With Freedom From Death and Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Death and Mitral Valve Surgery/Re-operation
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 133 | 73

140. Secondary Outcome: Number of Participants With Freedom From Death and Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Death and Mitral Valve Surgery/Re-operation
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 127 | 70

141. Secondary Outcome: Number of Participants With Freedom From Death and Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Death and Mitral Valve Surgery/Re-operation
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 122 | 66

142. Secondary Outcome: Number of Participants With Freedom From Death and Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Death and Mitral Valve Surgery/Re-operation
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 116 | 64

143. Secondary Outcome: Number of Participants With Freedom From Death and Mitral Valve Surgery/Re-operation
Description: Durability estimates: Freedom from Death and Mitral Valve Surgery/Re-operation
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 178 | 80
Participants | 111 | 61

144. Secondary Outcome: Number of Participants With MitraClip Device Embolization/Single Leaflet Device Attachment
Description: Device Embolization is defined as the complete detachment of the MitraClip Device from one or both mitral leaflets. Single leaflet device attachment (SLDA) is defined as attachment of one mitral valve leaflet to the MitraClip device. The control group did not receive the MitraClip device.
Time Frame: 12 months
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 0
Participants
  Device Embolization | 0 |
  Single Leaflet Device Attachment | 10 |

145. Secondary Outcome: Number of Participants With MitraClip Device Embolization/Single Leaflet Device Attachment
Description: as for outcome 144
Time Frame: 12 months to 3 years
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 0
Participants
  Device Embolization | 0 |
  Single Leaflet Device Attachment | 0 |

146. Secondary Outcome: Number of Participants With MitraClip Device Embolization/Single Leaflet Device Attachment
Description: as for outcome 144
Time Frame: 12 months to 4 years
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 0
Participants
  Device Embolization | 0 |
  Single Leaflet Device Attachment | 0 |

147. Secondary Outcome: Number of Participants With MitraClip Device Embolization/Single Leaflet Device Attachment
Description: as for outcome 144
Time Frame: 12 months to 5 years
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 0
Participants
  Device Embolization | 0 |
  Single Leaflet Device Attachment | 0 |

148. Secondary Outcome: Number of Participants With Non-cerebral Thromboembolism.
Description: Defined as any thrombus or thromboembolism in the vasculature (excluding central nervous system events) or on the investigational device or any commercially available implant used during surgery confirmed by standard clinical and laboratory testing and which requires treatment.
Time Frame: 12 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 3 | 3

149. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity of 0: None,1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe.
  "Discharge" refers to each individual patient's date of hospital discharge. The discharge date varies for each patient, but in general, discharge occurs before 30-days follow-up. A 30-day echocardiogram will be used if the discharge echocardiogram is unavailable or otherwise uninterpretable.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 173 | 76
Participants
  0: None | 2 | 16
  1+:Mild | 89 | 48
  2+: Moderate | 54 | 12
  3+: Moderate-to-Severe | 19 | 0
  4+: Severe | 9 | 0

150. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity of 0: None,1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 149 | 66
Participants
  0: None | 9 | 13
  1+:Mild | 55 | 38
  2+: Moderate | 57 | 14
  3+: Moderate-to-Severe | 21 | 1
  4+: Severe | 7 | 0

151. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity of 0: None,1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 127 | 57
Participants
  0: None | 2 | 3
  1+: Mild | 44 | 45
  2+: Moderate | 62 | 7
  3+: Moderate-to-Severe | 15 | 1
  4+: Severe | 4 | 1

152. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity of 0: None,1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 122 | 50
Participants
  0: None | 3 | 7
  1+:Mild | 45 | 36
  2+: Moderate | 55 | 5
  3+: Moderate-to-Severe | 19 | 2
  4+: Severe | 0 | 0

153. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity of 0: None,1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 105 | 49
Participants
  0: None | 4 | 4
  1+:Mild | 41 | 38
  2+: Moderate | 40 | 4
  3+: Moderate-to-Severe | 20 | 3
  4+: Severe | 0 | 0

154. Secondary Outcome: Number of Participants With MR Severity
Description: MR Severity of 0: None,1+: Mild, 2+: Moderate, 3+: Moderate-to-Severe, 4+: Severe
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 106 | 41
Participants
  0: None | 4 | 6
  1+:Mild | 49 | 32
  2+: Moderate | 34 | 2
  3+: Moderate-to-Severe | 18 | 1
  4+: Severe | 1 | 0

155. Secondary Outcome: Number of Participants With Non-cerebral Thromboembolism.
Description: as for outcome 148
Time Frame: 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 184 | 95
Participants | 1 | 2

156. Secondary Outcome: Number of Participants With Incidence of Mitral Valve Replacement
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 158 | 80
Participants | 17 | 11

157. Secondary Outcome: Number of Participants With Incidence of Mitral Valve Replacement
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
Number analyzed (Participants) | 167 | 84
Participants | 17 | 14

ADVERSE EVENTS:
Time Frame: 5 years
Description: The EVEREST II RCT enrolled 279 patients (184 Device and 95 Control), of whom 21 patients (6 Device and 15 Control) did not undergo treatment per their randomized assignment, and are reported as "randomized not treated" (RNT). Therefore, the Adverse Event was evaluated in 178 patients in Device group and 80 patients in Control group.
Arm/Group | Device Group (MitraClip Device) | Control Group (Mitral Valve Surgery)
All-Cause Mortality (participants affected / at risk) | 20/178 | 9/80
Serious Adverse Events (participants affected / at risk) | 127/178 | 54/80
Other Adverse Events (participants affected / at risk) | 168/178 | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Group (MitraClip Device) (N=178) | Control Group (Mitral Valve Surgery) (N=80)
Mitral Valve (MV) surgery (Cardiac disorders) | 1 (1) | 0 (0)
cardiac-single leaflet device attachment (SLDA) (Cardiac disorders) | 8 (9) | 0 (0)
Tamponade (Cardiac disorders) | 3 (3) | 0 (0)
Atrial arrhythmia (Cardiac disorders) | 30 (37) | 9 (12)
Atrial septal defect (Cardiac disorders) | 3 (3) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 6 (6) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (1)
Chest pain/angina (Cardiac disorders) | 9 (10) | 2 (2)
Congestive heart failure (Cardiac disorders) | 19 (31) | 10 (23)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Endocarditis (Cardiac disorders) | 3 (3) | 0 (0)
Heart block (Cardiac disorders) | 3 (3) | 2 (2)
Lead displacement (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve injury (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (4) | 0 (0)
Cardiac:Other (Cardiac disorders) | 3 (3) | 7 (7)
Cardiac:Other rhythm disorder (Cardiac disorders) | 7 (8) | 6 (6)
Pericardial effusion (Cardiac disorders) | 7 (7) | 4 (4)
Peripheral edema (Cardiac disorders) | 1 (1) | 0 (0)
Residual/recurrent mitral regurgitation (MR) (Cardiac disorders) | 21 (21) | 3 (3)
Supraventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Syncope/dizziness (Cardiac disorders) | 4 (6) | 1 (1)
Thrombus (Cardiac disorders) | 2 (3) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 7 (7) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 20 (20) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (3)
Gastro intestinal related:Bleed (Gastrointestinal disorders) | 10 (13) | 1 (1)
Gastro intestinal related:Infection (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastro intestinal related:Other (Gastrointestinal disorders) | 20 (24) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 16 (20) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Infection/bacteremia/septicemia (Blood and lymphatic system disorders) | 9 (10) | 2 (3)
Hematologic:Other (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 (11) | 5 (7)
Transient ischemic attack (TIA) (Nervous system disorders) | 7 (7) | 3 (3)
Intracerebral hemorrhage (Nervous system disorders) | 3 (3) | 1 (1)
Neurologic:Other (Nervous system disorders) | 5 (5) | 2 (2)
Neurologic:Stroke (Nervous system disorders) | 5 (5) | 3 (9)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Generalized weakness/fatigue:other (General disorders) | 3 (3) | 2 (2)
Infection:Other (Infections and infestations) | 4 (4) | 1 (1)
Mental disorders:Other (Psychiatric disorders) | 2 (2) | 0 (0)
Metabolic/endocrine disorders:Other (Metabolism and nutrition disorders) | 12 (12) | 6 (6)
Other (General disorders) | 23 (29) | 7 (10)
Fever (General disorders) | 0 (0) | 2 (2)
Incisional site pain (General disorders) | 0 (0) | 1 (1)
Skin/mucosal/subcutaneous tissue disorders:other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal-Infection (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal-Other (Renal and urinary disorders) | 3 (4) | 3 (3)
Renal insufficiency/failure (Renal and urinary disorders) | 12 (13) | 3 (3)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bronchial/lung disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory:Other (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 7 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 8 (8)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arteriovenous (AV) fistula (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (DVT) (Vascular disorders) | 5 (6) | 0 (0)
Peripheral Ischemia (Vascular disorders) | 1 (1) | 0 (0)
Bleeding complication (Vascular disorders) | 16 (17) | 5 (6)
Blood pressure complication (Vascular disorders) | 2 (2) | 0 (0)
Bruise/contusion/ecchymosis (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Hemodynamic instability (Vascular disorders) | 8 (8) | 2 (2)
Vascular:Injury (Vascular disorders) | 1 (1) | 1 (1)
Vascular:Other (Vascular disorders) | 3 (3) | 3 (3)
Pseudoaneurysm (Vascular disorders) | 3 (4) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 4 (4)
Vascular:Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Group (MitraClip Device) (N=178) | Control Group (Mitral Valve Surgery) (N=80)
Atrial arrhythmia (Cardiac disorders) | 23 (37) | 27 (33)
Bradyarrhythmia (Cardiac disorders) | 14 (16) | 6 (8)
Chest pain/angina (Cardiac disorders) | 33 (41) | 11 (14)
Congestive heart failure (Cardiac disorders) | 15 (22) | 11 (13)
Myocardial ischemia (Cardiac disorders) | 19 (21) | 6 (6)
Cardiac:Other rhythm disorder (Cardiac disorders) | 19 (21) | 11 (11)
Palpitations (Cardiac disorders) | 9 (9) | 5 (9)
Peripheral edema (Cardiac disorders) | 25 (28) | 23 (26)
Residual/recurrent mitral regurgitation (MR) (Cardiac disorders) | 29 (34) | 5 (5)
Syncope/dizziness (Cardiac disorders) | 38 (51) | 16 (18)
Ventricular arrhythmia (Cardiac disorders) | 9 (12) | 10 (12)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 5 (5)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 5 (5)
Cardiac:Other (Cardiac disorders) | 0 (0) | 12 (15)
Gastrointestinal:Other (Gastrointestinal disorders) | 79 (119) | 48 (81)
Gastrointestinal-Bleed (Gastrointestinal disorders) | 10 (13) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 32 (37) | 28 (32)
Hemolysis (Blood and lymphatic system disorders) | 11 (15) | 12 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13) | 7 (7)
Hematologic:Other (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Connective tissue disorders:other (Musculoskeletal and connective tissue disorders) | 76 (114) | 26 (44)
Transient ischemic attack (TIA) (Nervous system disorders) | 11 (12) | 9 (10)
Neurologic:Other (Nervous system disorders) | 16 (21) | 14 (17)
Fever (General disorders) | 17 (19) | 13 (14)
Generalized weakness/fatigue (General disorders) | 32 (43) | 25 (30)
Incisional site pain (General disorders) | 49 (60) | 49 (53)
Mental disorders:other (Psychiatric disorders) | 28 (35) | 25 (32)
Metabolic/endocrine disorders:other (Metabolism and nutrition disorders) | 49 (73) | 38 (58)
Other (General disorders) | 78 (133) | 35 (60)
Skin/mucosal/subcutaneous tissue disorders:other (Skin and subcutaneous tissue disorders) | 14 (19) | 5 (7)
Renal:Infection (Renal and urinary disorders) | 10 (16) | 9 (12)
Renal-Other (Renal and urinary disorders) | 19 (22) | 6 (6)
Renal insufficiency/failure (Renal and urinary disorders) | 10 (15) | 9 (11)
Bronchial/lung disorders (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 22 (24)
Respiratory:Infection (Respiratory, thoracic and mediastinal disorders) | 18 (22) | 10 (11)
Respiratory:Other (Respiratory, thoracic and mediastinal disorders) | 79 (115) | 30 (45)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 27 (31)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Bleeding complication (Vascular disorders) | 62 (73) | 17 (18)
Blood pressure complication (Vascular disorders) | 19 (23) | 14 (18)
Bruise/contusion/ecchymosis (Vascular disorders) | 26 (32) | 5 (5)
Hematoma (Vascular disorders) | 26 (29) | 0 (0)
Hemodynamic instability (Vascular disorders) | 45 (55) | 27 (31)
Vascular:Other (Vascular disorders) | 9 (11) | 0 (0)
Blood transfusion (Vascular disorders) | 0 (0) | 8 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
mitral stenosis (Cardiac disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days